CLINICAL TRIAL: NCT04302155
Title: Wii Fit as Balance Assessment and Training Tool for Young Adults
Brief Title: Wii Fit as Balance Assessment and Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Aruba Saeed REC/00216
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Healthy Young Adults
Keywords: Wii Fit; Balance Training; Young Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nintendo Wii (Experimental): Balance-specific exer-games focusing on dynamic aspects of center of pressure (COP) on Wii fit system.
  Interventions: Other: balance-specific -games focusing on dynamic aspects of COP on Wii fit system.
- Traditional (Experimental): Mini trampoline two balance exercises of 6 minutes on mini trampoline for a total duration of 3 min on each leg Inflatable discs 4 balance exercises of 12 minutes on BOSU ball 6 minutes on rounded side and 6 minutes on rigid side.
  Interventions: Other: mini trampoline and inflatable discs group

INTERVENTIONS:
Other: balance-specific -games focusing on dynamic aspects of COP on Wii fit system. — The participants were randomly assigned into two groups interventional and control. Total 18 minutes session was given to both groups wii fit group and traditional balance training group. All participants were given 3 sessions per week for 6.
  Total 48 participants were initially accessed initially for eligibility , 13 participants were excluded because of having good balance and good balance age score on Wii fit assessment, 35 participants were recruited for balance training. These participants were randomly divided into Wii fit and traditional training group through sealed enveloped method 18 participants was recruited in Wii fit group and 17 in traditional balance training group. 3 participants drop out from Wii fit group and 2 from traditional balance training group.
  Some examples include catching apples in a basket ,moving a golf ball around barriers towards a hole , popping rising balloons/bubbles and air hockey .
  Arms: Nintendo Wii
Other: mini trampoline and inflatable discs group — High skipping and landing on a limb every time (2 repeats of 45 s each leg).Standing on one leg and try to catch the ball thrown at them in various directions by the researcher (2 repeats of 45 s each leg) Exercises in inFlated rubber hemisphere attached toa rigid platform (BOSU)
  1. Standing on BOSU's round soft surface with one foot, in an attempt to maintain balance (2 repeats of 45 s each leg).
  2. Standing on BOSU's round soft surface with one foot, in an attempt to maintain balance, while lifting the non-support leg forward and backward (2 repeats of 45 s each leg).
  3. Standing on BOSU flat hard surface with both legs, in an attempt to maintain balance (3 minutes on both legs).
  4. Standing on BOSUs flat hard surface with both feet, in an attempt to maintain balance, while trying to catch the ball thrown at them by the experimenter in various directions (3 minutes on both leg)
  Arms: Traditional

SUMMARY:
Balance play a vital role to increase motor skills in healthy young adults. With increasing age balance control ability decreases,this decline can result as early as mid-30s. In young adults focus on improving anticipatory postural control so risk of lower extremity injuries especially ankle and knee injuries can be minimized and future risk of fall can be minimized.Objective is To compare the effect of traditional versus Wii fit training on balance in young adults the participants were randomly assigned into two groups interventional and control. total 18 minutes session was given to both groups wii fit group and traditional balance training group. all participants were given 3 sessions per week for 6. participants were initially accessed initially for eligibility , these participants were randomly divided into wii fit and traditional training group through sealed enveloped method . the initial assessment was done on wii fit. balance intervention to wii fit group is different games available on wii fit software. balance intervention given to traditional group is on trampoline and on BOSU ball.

DETAILED DESCRIPTION:
Balance is an integral part of human ability. Whether for daily activities in life or sports related activities, humans rely on body balance and it affects peoples successful performance.To maintain balance, individuals must control their center of mass (COM) location over the base of support (BOS) during both voluntary movements, and in response to external, destabilizing forces. Exercises play an important role in balance improvement and fall prevention. Physiotherapists can help individuals to train their central nervous system to respond to different sensory challenges through balance control exercises. Falls are a leading public health concern with statistics reporting that 30 percent of adults 65 years of age and older, and 50 per cent of those 80 years of age and older, experience a fall annually. Research highlights the importance of patient-orientated, balance-targeted exercises, which draw focus to a sense of body position in space. virtual reality and video gaming programs for improving balance. An increasingly popular system for virtual reality balance training is the Nintendo Wii. Nintendo Wii real-time device is somatosensory gaming comprises the balance board, software, and database it is used for balance assessment are balance training purpose. Virtual reality balance training typically requires participants to produce discrete, controlled movements to and beyond their base of support in response to visual targets. A force plate measures the performance of the participant and can provide online feedback of postural control.

Literature shows its high levels of usability and enjoyment with no serious adverse effects. Findings of research on effects of the Nintendo Wii Fit on Community-Dwelling Adults with Perceived Balance Deficits suggest that an intervention program including the Wii fit may be an effective rehabilitation option for adults with perceived balance deficits.

The advantage of the Nintendo Wii with Wii Balance Board (WBB) is that it not only offers an alternative balance exercise-training tool but it can also record balance measurements. The WBB is more portable than heavy and expensive laboratory equipment while still providing valid and reliable measurements. A recent study evaluated the validity of the WBB in measuring balance variables.There are number of exercise training that are used for balance improvement including tai chi, yoga , task specific training. Some of them showed marked improvement in balance while others have little or no improvement. The use of exergaming for different types of rehabilitation has established great interest particularly Nintendo Wii .Wii fit is has been used for balance training from the past few years in an individual with balance impairment as well as in healthy individuals, it is a novel and in expansive method of balance training in WBB use improve the visual perception, postural control, mobility, motor function and also decrease the risk of fall . Different games are used in WBB including Balance training, Yoga, strength training, aerobic training. Few studies used the control group along with Wii fit group to determine its effectiveness in balance training. Different clinical test for balance assessment was used before and after balance training including Berg Balance Scale (BBS), Fullerton Advance Balance test(FAB) test, Time up and go test (TUG), Functional Reach Test (FR) in different studies.A study showed that balance interventions involving the Wii Fit system have relied on the balance-specific exer-games it involve Wii Fit balance games, yoga games rely on static balance control. Despite this broad mission, the Wii Fit has generated specific interest in the domain of neurorehabilitation as a measurement and training device for balance ability. Balance control increases with increasing age as early as mid-30s .Balance control increases with increasing age as early as mid-30s This study aimed to assess the balance error in healthy young adults of our society as well as their balance training by using Wii fit and traditional balance training. By providing balance training to young population we intended to improve feed forward postural control, improve motor skills and decrease chances of lower extremity injuries

ELIGIBILITY:
Inclusion Criteria:

* Healthy young adults (18 to 30 years)
* Either gender
* having static standing balance of 30 seconds with eye open and eye close.
* Willing to participate
* Normal or corrected vision and hearing, no history of primary medical risk factors for falls
* Adults having wii fit balance age greater > years from their actual age

Exclusion Criteria:

* Young adults with any diagnosed balance issue
* Young adults with pathology of the musculoskeletal, neurological or vestibular system, severe cardiovascular disease, diabetes, adults using beta-blockers or antidepressants.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2018-08-15 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2019-01-15 (Actual)

PRIMARY OUTCOMES:
Fullerton advance balance test (FAB) | 4 weeks
  As per baseline assessment.This test is basically used to identify the balance problem in active adults. This test is used for the assessment of static and dynamic balance assessment under different situations. It include 10 activities, its total score is 40 cut off score is 25. >25 means risk of fall absent. <25 means risk of fall present. Its test retest reliability is (ICC=0.98)
  Components of FAB:
  * Stand with feet together and eyes closed
  * Reach forward to retrieve an object (pencil) held at shoulder height with outstretched arm
  * Turn 360 degrees in right and left directions
  * Step up onto and over a 6-inch bench
  * Tandem walk
  * Stand on one leg
  * Stand on foam with eyes closed
  * Two-footed jump
  * Walk with head turns
  * Reactive postural control
Y balance test: | 4 weeks
  As per baseline assessment.Y-Balance Test is reliable tool for balance assessment. The person stand on one leg and simultaneously reaches other leg far in three directions:anterior, posterolateral, posteromedial. It measures muscle's flexibility, strength and balance
Wii fit system | 4 weeks
  As per baseline assessment. Wii fit is also used for static and dynamic center of pressure control. According to dynamic center of pressure variation from midline during performing different task Wii fit age is calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Arshad Nawaz Malik, PHD, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pompeu JE, Mendes FA, Silva KG, Lobo AM, Oliveira Tde P, Zomignani AP, Piemonte ME. Effect of Nintendo Wii-based motor and cognitive training on activities of daily living in patients with Parkinson's disease: a randomised clinical trial. Physiotherapy. 2012 Sep;98(3):196-204. doi: 10.1016/j.physio.2012.06.004. Epub 2012 Jul 25. PMID 22898575
- [Background] Chang WD, Chang WY, Lee CL, Feng CY. Validity and reliability of wii fit balance board for the assessment of balance of healthy young adults and the elderly. J Phys Ther Sci. 2013 Oct;25(10):1251-3. doi: 10.1589/jpts.25.1251. Epub 2013 Nov 20. PMID 24259769
- [Background] Whyatt C, Merriman NA, Young WR, Newell FN, Craig C. A Wii Bit of Fun: A Novel Platform to Deliver Effective Balance Training to Older Adults. Games Health J. 2015 Dec;4(6):423-33. doi: 10.1089/g4h.2015.0006. Epub 2015 Oct 15. PMID 26469308
- [Background] Lange B, Chang CY, Suma E, Newman B, Rizzo AS, Bolas M. Development and evaluation of low cost game-based balance rehabilitation tool using the Microsoft Kinect sensor. Annu Int Conf IEEE Eng Med Biol Soc. 2011;2011:1831-4. doi: 10.1109/IEMBS.2011.6090521. PMID 22254685
- [Background] Goble DJ, Cone BL, Fling BW. Using the Wii Fit as a tool for balance assessment and neurorehabilitation: the first half decade of "Wii-search". J Neuroeng Rehabil. 2014 Feb 8;11:12. doi: 10.1186/1743-0003-11-12. PMID 24507245
- [Background] Meldrum D, Glennon A, Herdman S, Murray D, McConn-Walsh R. Virtual reality rehabilitation of balance: assessment of the usability of the Nintendo Wii((R)) Fit Plus. Disabil Rehabil Assist Technol. 2012 May;7(3):205-10. doi: 10.3109/17483107.2011.616922. Epub 2011 Nov 25. PMID 22117107
- [Background] Franco JR, Jacobs K, Inzerillo C, Kluzik J. The effect of the Nintendo Wii Fit and exercise in improving balance and quality of life in community dwelling elders. Technol Health Care. 2012;20(2):95-115. doi: 10.3233/THC-2011-0661. PMID 22508022